CLINICAL TRIAL: NCT05279482
Title: Comparison Between Standard Dose Methyl Prednisolone and Megadose Methyl Prednisolone as Regards Outcome in SARS.COV.2 Patients in Intensive Care Unit : Retrospective Study
Brief Title: Comparison Between Different Doses of Steroids in COVID-19 Patients
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr M Hilal Abdou, Assistant Professor, Ain Shams University
Other Study IDs: MS41/2022
Record Dates: First submitted 2022-03-10; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness; Pneumonia, Viral
MeSH Terms: conditions — Critical Illness; Pneumonia, Viral | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group treated with standard dose methyl prednisolone: patients with positive PCR and requiring oxygen therapy
  Interventions: Other: observation for outcome of methylprednisolone dose
- group treated with mega dose methyl prednisolone: patients with positive PCR and requiring oxygen therapy
  Interventions: Other: observation for outcome of methylprednisolone dose

INTERVENTIONS:
Other: observation for outcome of methylprednisolone dose — no intervention as it is retrospective study for outcome

SUMMARY:
aim of this study is to compare between standard dose methyl prednisolone and mega dose methyl prednisolone as regards outcome reflected by mortality rate, percentage of mechanically ventilated patients and icu length of stay of covid 19 patients admitted in intensive care unit.

DETAILED DESCRIPTION:
Retrospective study for comparison between standard dose methyl prednisolone and mega dose methyl prednisolone as regards outcome reflected by mortality rate ,percentage of mechanically ventilated patients and icu length of stay of covid 19 patients admitted in intensive care unit.

Previous studies suggested that cytokine release syndrome could be involved in the pathophysiology of critical SARS.COV.2 resulting in death so early suppression of cytokine storm may be lifesaving in critical patients.

ELIGIBILITY:
Inclusion Criteria:

* All icu admitted covid 19 patients with positive PCR, diagnosed by CT chest and needing oxygen therapy

Exclusion Criteria:

* Not requiring oxygen therapy
* Negative PCR
* Uncontrolled blood sugar or DKA
* Patients on long term steroids therapy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: SARS.COV.2. admitted in intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
28 days mortality rate | 1 month
  observation for mortality rate in both groups

SECONDARY OUTCOMES:
mechanical ventilation and icu length of stay | up to 3 months
  observation for percentage of mechanically ventilated patients and length of stay

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ain shams university hospitals, Cairo
  - Faculty of medicine, Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: Undecided